CLINICAL TRIAL: NCT01323608
Title: The Effect of Vitamin D Supplementation on Calcium Excretion in Thalassemia: a Dose Response Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Maria Vogiatzi, MD, Weill Cornell Medical College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1102011521
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Thalassemia Major
Keywords: Thalassemia; hypercalciuria; vitamin D; To conduct a pilot study to determine the effect of various doses of; vitamin D supplementation on vitamin D stores and their association with calcium excretion
MeSH Terms: conditions — beta-Thalassemia; Thalassemia; Hypercalciuria | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Low Vitamin D Group (Experimental): Subjects in this group will receive the equivalent of 400 IU/day.
  Interventions: Drug: Vitamin D3
- Intermediate Vitamin D group (Experimental)
  Interventions: Drug: Vitamin D3
- High Vitamin D Group (Experimental)
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D3 will be given at the equivalent of the following doses: 400, 1000, and 2000 IU/day.
  Arms: High Vitamin D Group; Intermediate Vitamin D group; Low Vitamin D Group
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this pilot study is to determine the effect of various doses of vitamin D supplementation on vitamin D stores and calcium excretion in the urine in subjects with Thalassemia Major (TM). Subjects with TM are routinely placed on vitamin D supplements because they frequently have osteoporosis (a condition in which bone tissue thins and loses density and strength) and low vitamin D stores. The amount of vitamin D supplementation that is required to raise vitamin D stores in optimal levels is not known in TM, and will be determined in this study. Finally, a recent study in TM has linked blood vitamin D levels to urine calcium excretion, which is a risk factor for kidney stones. Therefore, we want to determine changes in calcium excretion with various vitamin D doses and with increasing vitamin D stores. We plan to test 3 doses of vitamin D for 3 months in children and adults with TM. Changes in vitamin D blood levels and urinary calcium will be determined. The results of this pilot study will be used in future studies that will examine the effect of various doses of vitamin D supplementation in the treatment of osteoporosis in TM.

DETAILED DESCRIPTION:
Specific Aim: To determine the effect of various doses of vitamin D supplementation on serum concentration of 25 hydroxy vitamin D (25OHD) and urinary calcium excretion in adults and children with TM.

Hypothesis: Vitamin D supplementation at doses that result in serum 25OHD levels >30 ng/ml result in high rates of hypercalciuria (i.e. increased urinary calcium excretion) in children and adults with TM.

The pilot study will be performed at Weill Cornell Medical College, Payson 695.

* Children and adults with TM, will be divided into 4 groups: "standard" vitamin D dose (equivalent to 400 IU/day), "intermediate" vitamin D dose (equivalent to 1000 IU/day), "high" vitamin D dose (equivalent to 2,000 IU/day) and a "placebo" group that will receive an inactive ingredient. 10 subjects will be assigned to each group. The duration of the study will be 3 months.
* While some studies found no difference between vitamin D2 and D3, others suggest that vitamin D3 may be more advantageous in restoring 25 OHD concentrations. For these reasons, vitamin D3 will be used in this protocol.
* Study schedule with study interventions and frequencies is set out below (see table). All 4 groups will adhere to the same schedule. After obtaining consent, subjects will have a "Baseline Visit", which will include: 1) a complete physical examination; 2) laboratory evaluation that includes measurement of 25OHD, which is the major circulating form of vitamin D and reflects the body's vitamin D stores. Additional blood and urine samples will be obtained for measurement of urinary calcium excretion and serum Calcium and parathyroid hormone (PTH); and 3) Dietary calcium intake questionnaire. 4) Start of study medication.
* Subjects will then return every 2-4 weeks for routine blood transfusions and as required for the management of Thalassemia. To ensure compliance, study medications will be administered by study personnel during these routine visits. Vitamin D supplies will be packaged according to one week worth requirement, i.e. as 1,000 IU/day x 7days=7,000 IU for the "intermediate" vitamin D group. The dose that will be administered during these visits will depend on the interval between transfusions, i.e. 7,000 IU x 2weeks, for a subject of the "intermediate" dose who is transfused every two weeks.
* At the end of 3 month treatment, subjects will have a final visit, that is also scheduled to coincide with a routine transfusion visit. Subjects will have the same evaluation and procedures as in "Baseline Visit" : 1) a complete physical examination; 2) fasting laboratory evaluation that includes measurement of 25OHD, urinary calcium excretion and serum Calcium and PTH; and 3) Dietary calcium intake questionnaire.
* Subjects will be asked to take calcium supplementation at the dose of 500 mg daily for the 6-8 year old and 1,000 mg daily for the 9-18 year old subjects. This intervention will ensure adequate calcium intake in both groups.

All labs will be processed at the CTSC Core Lab. Study meds will be distributed by the central pharmacy. Investigational drug will be administered by study personnel during the transfusion visits to ensure compliance.

Eligible subjects will be assigned to a study group following a block type of enrollment. To ensure an equal, or near equal sex and age distribution, study groups will be matched according to sex and age. Half of the subjects in each group will be composed of pediatric subjects and the other half will be composed of adult subjects.

Study Schedule and Procedures:

* Baseline visit: Physical Exam, 25OHD, Intact PTH & Serum Calcium, 24 hr & spot urine collection for Ca/Crea, Calcium intake questionnaire, Vitamin D Supplementation/Placebo.
* Every 2-4 weeks: Administration of Vitamin D/Placebo
* 3 Month Visit: Physical Exam, 25OHD, Intact PTH & Serum Calcium, 24 hr & spot urine collection for Ca/Crea, Calcium intake questionnaire, and Vitamin D Supplementation/ Placebo.

Primary study endpoint:

Changes in 25OHD concentrations and calcium excretion with the various vitamin D3 doses will be determined at the end of the study and constitute the primary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Thalassemia Major (TM)
* 25 OHD: 15-29 ng/ml
* Age 6 to 60 years
* Albumin corrected serum Calcium: Normal (8.5-10.5 mg/dl)

Exclusion Criteria:

* Other thalassemia syndromes
* 25 OHD concentrations < 15 ng/ml or ≥30 ng/ml
* Subjects younger than 6 years
* Hypoparathyroidism
* Abnormal albumin corrected serum Ca (i.e. total calcium <8.5 or > 10.5 mg/dl)
* Medications that may adversely affect vitamin D metabolism (anticonvulsants) or absorption
* End stage renal, heart, or liver disease
* History of Nephrolithiasis or Nephrocalcinosis
* Diseases associated with hypercalciuria (ie. Sarcoidosis, Cushing syndrome, and Wilson disease to name a few)

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Vitamin D Dose Response Curve | 3 Months
  To perform a dose response curve for vitamin D supplementation study and determine the relationship between vitamin D doses and serum 25OHD concentrations and urinary calcium excretion in children and adults with TM.

SECONDARY OUTCOMES:
Vitamin D Dose Response Curve | 3 Months
  To determine changes in serum calcium and PTH concentrations with various vitamin D doses

CONTACTS AND LOCATIONS:
Overall Officials: Maria Vogiatzi, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States